CLINICAL TRIAL: NCT04928807
Title: A Multicenter, Randomized, Open-label, Controlled Phase III Clinical Trial of Short-Course Radiotherapy Followed by Neoadjuvant Chemotherapy and Camrelizumab in the Treatment for Locally Advanced Rectal Cancer
Brief Title: Short-Course Radiotherapy Followed by Neoadjuvant Chemotherapy and Camrelizumab in Locally Advanced Rectal Cancer (UNION)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Tao Zhang, Chief of gastrointestinal oncology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-CRC-Ⅲ-006
Record Dates: First submitted 2021-06-14; First posted 2021-06-16 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short course radiotherapy sequential camrelizumab and chemotherapy (Experimental): Radiotherapy will employ conformal or intensity-modulated radiation therapy, with a pelvic irradiation dose of 25 Gy/5 Fractions/1 week. Then rest for 1 week after radiotherapy and begin to receive neoadjuvant chemotherapy CAPOX and camrelizumab, for 2 cycles.
  The patients were operated within 10 weeks after the last radiotherapy, and the surgical method is total mesorectal excision.
  Postoperative adjuvant therapy will be started 4-6 weeks after surgery, and the adjuvant regimen was the same as that before operation (CAPOX + camrelizumab) for 6 cycles
  Interventions: Combination Product: Short course radiotherapy sequential camrelizumab and chemotherapy
- Long term concurrent chemoradiotherapy and sequential chemotherapy (Active Comparator): The patients received neoadjuvant therapy of CAPOX 2 weeks after long-term concurrent chemoradiotherapy (28*1.8Gy, during the same period, capecitabine was 825 mg / m2, twice a day, 5 days a week).
  The patients were operated within 10 weeks after the last radiotherapy. Adjuvant therapy should begin within 4-6 weeks after surgery, and the adjuvant regimen was the same as that before operation (CAPOX) for 6 cycles
  Interventions: Combination Product: Short course radiotherapy sequential camrelizumab and chemotherapy

INTERVENTIONS:
Combination Product: Short course radiotherapy sequential camrelizumab and chemotherapy — Short course radiotherapy, 5 * 5Gy, once a day, 5Gy each time, for 5 days, continuous irradiation, three-dimensional 3D-CRT or IMRT technology is recommended camrelizumab 200 mg , D1, intravenous drip, q3w, 2 cycles before operation, postoperative adjuvant treatment, the longest medication time of camrelizumab was less than 1 year during the whole study period; Capecitabine 1000 mg / m2, twice a day, oral, 1-14 days, then rest for 7 days, q3w, 2 cycles before operation and 6 cycles after operation; Oxaliplatin 130 mg / m2, D1, intravenous infusion 2 hours, q3w, 2 cycles before operation, 6 cycles after operation

SUMMARY:
The study is a multicenter, open-label, randomized controlled clinical study, and the purpose of the study is to compare the pathological complete response rate (PCR) of patients with locally advanced rectal cancer treated with short-term radiotherapy, sequential Camrelizumab and CAPOX (group A) to long-term concurrent chemoradiotherapy, sequential CAPOX (group B) in patients with LARC. A total of 230 patients were included in this study.

DETAILED DESCRIPTION:
Patients with locally advanced rectal cancer (T3-4/N+) were randomly assigned to experimental group A or control group B according to the ratio of 1:1,who will receive preoperative neoadjuvant therapy, and the Primary endpoint of the study is Pathological complete response rate(PCR ) assessed by the blind independent review committee (BIRC), defined as the absence of viable tumour cells in the resected primary tumour specimen and all sampled regional lymph nodes (ypT0N0)

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their family members agree to participate in the study and sign the informed consent form;
2. Age 18-75 years, male or female;
3. Histologically confirmed T3-44 and/or N+ rectal adenocarcinoma (AJCC/UICC TNM staging (8th Edition, 2017);
4. inferior margin ≤ 10 cm from the anal verge;
5. It is expected to reach R0;
6. ECOG performance status score is 0-1;
7. Swallowing pills normally;
8. Untreated with anti-tumor therapy for rectal cancer, including radiotherapy, chemotherapy, surgery, etc;
9. Surgical treatment is planned after neoadjuvant treatment;
10. There was no operative contraindication;
11. Laboratory tests were required to meet the following requirements:

    white blood cell (WBC) ≥ 4×109/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet count ≥ 100×109/L; Hemoglobin ≥90 g/L; Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN); Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Serum creatinine ≤1.5 times the upper limit of normal value or creatinine clearance rate ≥50 mL/min; International normalized ratio (INR) ≤ 1.5 × ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN
12. Males or females with reproductive ability who are willing to use contraception in the trial;

Exclusion Criteria:

1. Documented history of allergy to study drugs, including any component of Camrelizumab, capecitabine, irinotecan, oxaliplatin and other platinum drugs;
2. Have received or are receiving any of the following treatments:

   Any radiotherapy, chemotherapy or other anti-tumor drugs for tumor; Patients who need to be treated with corticosteroid (dose equivalent to prednisone of >10 mg/day) or other immunosuppressive agents within 2 weeks prior to study drug administration; Received live attenuated vaccine within 4 weeks before the first use of the study drug; Major surgery or severe trauma within 4 weeks before the first use of the study drug;
3. Any active autoimmune disease or history of autoimmune disease;
4. Have a history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation or allogeneic bone marrow transplantation;
5. There are clinical symptoms or diseases of heart that are not well controlled;
6. Severe infection (CTCAE > 2) occurred within 4 weeks before the first use of the study drug; Baseline chest imaging revealed active pulmonary inflammation, signs and symptoms of infection within 14 days prior to the first use of the study drug, or oral or intravenous antibiotic therapy, except for prophylactic use of antibiotics;
7. Patients with active pulmonary tuberculosis infection found by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within one year before enrollment, or with a history of active pulmonary tuberculosis infection more than one year ago but without regular treatment;
8. The presence of active hepatitis B (HBV DNA > 2000 IU/mL or 104 copies/mL) was positive for hepatitis C (hepatitis C antibody) and HCV RNA was higher than the lower limit of analytical method;
9. Female subject who is pregnant or breastfeeding;
10. Patients who are not suitable for participation in clinical trials in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) rate | an expected average of 5 months
  Pathological complete response rate (PCR) assessed by the blind Independent Review Committee, defined as the absence of viable tumour cells in the resected primary tumour specimen and all sampled regional lymph nodes (ypT0N0)

SECONDARY OUTCOMES:
3-year event-free survival rate | an expected average of 3 years
  The percentage of patients without disease recurrence or progression or death due to any cause after 3-year follow-up
Overall Survival | an expected average of 5 years
  The time from the date of randomization to the death caused by any cause
R0 resection rate | an expected average of 2 years
  The rate of negative margin microscopically
3-year disease-Free Survival | an expected average of 3 years
  The time from the first day of disease free (operation date) to local or distant recurrence, or the death event caused by any reason, whichever occurs first
dverse events (AEs) were graded according to the NCI CTCAE version 5·0 | an expected average of 1.5 years
  Adverse events and surgical safety

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zhang F, Yu D, Yang J, Zhai M, Li L, Zhao L, Wang J, Zhang T, Lin Z. Pretreatment high cholesterol and low neutrophils predict complete pathological response after neoadjuvant short-course radiotherapy followed by chemotherapy and immunotherapy in locally advanced rectal cancer. Oncol Lett. 2023 Jun 7;26(1):319. doi: 10.3892/ol.2023.13905. eCollection 2023 Jul. PMID 37332340